CLINICAL TRIAL: NCT04762706
Title: Treating the Whole Patient: Measuring Distress in Prosthetic Joint Infection Using a Standardized Metric: CRUTCH Pathway Pilot.
Brief Title: Measuring Distress in Prosthetic Joint Infection Using a Standardized Metric: CRUTCH Pathway Pilot.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Allison Lastinger, Assistant Professor, West Virginia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2101221058
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Prosthetic Joint Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CRUTCH Pathway (Experimental): A novel behavioral health program.
  Interventions: Behavioral: CRUTCH Pathway

INTERVENTIONS:
Behavioral: CRUTCH Pathway — Patients will be offered referral to a behavioral medicine specialist in the novel Combined Rehabilitation Using Team Centered Help (CRUTCH) Pathway. Once enrolled, these patients will meet virtually with a psychiatrist. The psychiatrist will complete a 30-minute intake visit where he will review the patient's DT scoring, discuss contributing factors to current distress level, and assess for psychiatric comorbidities. Following this assessment, psychotherapy, psychotropic medication, and referral for social work/financial services will be offered to the patient as indicated. If more frequent behavioral health follow-up is clinically indicated, it will be provided to the patients.

SUMMARY:
The purpose of this study is to determine whether patients being treated for prosthetic joint infections (PJI) experience distress during the course of their treatment and how distress influences various aspects of their lives. WVU expects to enroll approximately 12 subjects. Patients identified as scoring ≥4 on the Distress Thermometer at the two-week follow-up visit will be offered the opportunity to participate in the novel CRUTCH Pathway. Once enrolled, you will meet virtually with a mental health provider. The mental health provider will complete a 30-minute intake visit where he will review your distress thermometer scoring, discuss contributing factors to current distress level, and assess for psychiatric comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* ability to speak and read English, and cognitively sound. Patients scheduled for revision of total hip or knee arthroplasty will be categorized as septic or aseptic revisions. Patients identified as scoring ≥4 on the DT at the two-week follow-up visit.

Exclusion Criteria:

* Patients younger than 18 or older than 89, patients unable to speak and/or read English, and patients who are not able to understand and answer questions asked on surveys. Elective primary total hip or knee arthroplasty, hemiarthroplasty, unicompartmental knee arthroplasty.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Assess patient experience with a Distress Thermometer and Problem List | Two week post operative
  Distress Thermometer and Problem List for Patients with a score from 0-10, where 0 is no distress and 10 extreme distress.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Lastinger, MD, Principal Investigator — West Virginia University
Locations (1):
- WVU Medicine University Town Center, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT04762706/ICF_000.pdf